CLINICAL TRIAL: NCT03311919
Title: Exploratory Study of "Natural Killer" Inflammatory Lymphocytes in Waste Per-operating of Tonsillectomy
Acronym: LINK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/204
Record Dates: First submitted 2017-09-27; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Tonsillectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to describe the frequency of the presence of cells Natural Killer (NK) expressing CD86 and HLA - DR in tonsils

ELIGIBILITY:
Inclusion Criteria:

* patient with programmed tonsillectomy as part of the care

Exclusion Criteria:

* patient opposition to use its waste of per-operating tonsillectomy for research purposes
* patient with immunosuppressive and/or corticoid treatment (> 1 mg/kg)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with tonsillectomy
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
presence of lymphocytes NK expressing CD86 and HLA - DR | inclusion
  by immunostaining and detection by flow cytometry

REFERENCES:
- [Background] Loyon R, Picard E, Mauvais O, Queiroz L, Mougey V, Pallandre JR, Galaine J, Mercier-Letondal P, Kellerman G, Chaput N, Wijdenes J, Adotevi O, Ferrand C, Romero P, Godet Y, Borg C. IL-21-Induced MHC Class II+ NK Cells Promote the Expansion of Human Uncommitted CD4+ Central Memory T Cells in a Macrophage Migration Inhibitory Factor-Dependent Manner. J Immunol. 2016 Jul 1;197(1):85-96. doi: 10.4049/jimmunol.1501147. Epub 2016 May 27. PMID 27233967